CLINICAL TRIAL: NCT01983709
Title: A Phase 1 Study of Allogeneic Human Bone Marrow Derived Mesenchymal Stem Cells in Localized Prostate Cancer
Brief Title: Allogeneic Human Bone Marrow Derived Mesenchymal Stem Cells in Localized Prostate Cancer
Acronym: MSC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was Terminated by PI due to low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1348; NA_00083720 (Other: JHMIRB)
Record Dates: First submitted 2013-10-28; First posted 2013-11-14 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Human Mesenchymal Stem Cells (Experimental): This will be a dose escalation study. The first 3 subjects will receive a single dose of 1 x 10^6 cells/kg or a maximum dose of 1 x 10^8 total cells IV.
  The remaining subjects will receive a single dose of 2 x 10^6 cells/kg or a maximum dose of 2 x 10^8 total cells IV.
  Interventions: Biological: Allogeneic Human Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Allogeneic Human Mesenchymal Stem Cells — This will be a dose escalation study. The first 3 subjects will receive a single dose of 1 x 10^6 cells/kg or a maximum dose of 1 x 10^8 total cells IV 4 days prior to undergoing a planned prostatectomy.
  The remaining subjects will receive a single dose of 2 x 10^6 cells/kg or a maximum dose of 2 x 10^8 total cells IV either 4 or 6 days prior to the planned prostatectomy, and if additional doses of MSCs are able to be expanded, up to 6 additional men will be enrolled with a plan to treat them 8 days prior to the prostatectomy.

SUMMARY:
The objective of this study is to determine if systemically infused allogeneic bone marrow derived mesenchymal stem cells (MSC) home to sites of prostate cancer in men with localized adenocarcinoma of the prostate that are planning to undergo a prostatectomy. Investigators plan to systemically infuse MSCs 4, 6 or 8 days prior to enrolled subjects' planned prostatectomies. Investigators will then quantify the relative amount of donor MSC DNA to recipient DNA present in patients' explanted prostate specimens. This will be accomplished via BEAMing digital PCR. This trial will provide the foundation for future studies aimed at engineering MSCs to deliver a toxin to sites of metastatic prostate cancer.

ELIGIBILITY:
MSC Donors

Inclusion Criteria:(MSC donor cohort):

1. Age ≥18 years, ≤30 years
2. Male sex
3. Donor must meet the selection and eligibility criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT) and FDA 21 CFR Part 1271

Exclusion Criteria:(MSC donor cohort):

1. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
2. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
3. Inability to provide informed consent.

MSC Recipients

Inclusion Criteria (Treatment cohort):

1. Age ≥18 years
2. Eastern cooperative group (ECOG) performance status ≤2
3. Documented histologically confirmed adenocarcinoma of the prostate
4. Gleason score on diagnostic biopsy specimens of ≥ 6
5. ≥ 3 positive cores within diagnostic biopsy specimens
6. At least one prostate core must contain ≥ 30% prostate cancer
7. Scheduled to undergo a prostatectomy at Johns Hopkins
8. Has not received systemic therapy for prostate cancer (i.e. LHRH agonist/antagonist therapy)
9. Sexual Health Inventory in Men (SHIM) score ≥ 17

Exclusion Criteria (Treatment cohort):

1. Prior radiation therapy to the prostate.
2. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
3. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
4. Inability to provide informed consent.
5. Any active autoimmune disease requiring treatment (e.g. steroid, disease-modifying antirheumatic drugs, biologic agents, etc.).
6. Prior history of penicillin or streptomycin allergy.
7. No prior history of deep venous thrombosis or pulmonary embolism within 5 years prior to enrollment in the study.
8. Abnormal liver function (bilirubin, AST, ALT ≥ 3 x upper limit of normal)
9. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
10. Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within the last five years prior to enrollment in the study.
11. History of symptomatic pulmonary dysfunction.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Amount of systemically infused (MSC) DNA relative to recipient DNA at sites of prostate cancer in men with localized adenocarcinoma of the prostate that are scheduled to undergo a prostatectomy | Up to 3 years
  Allogeneic MSCs will be quantified through tissue BEAMing and the percent of MSCs per total cell number will be calculated.

SECONDARY OUTCOMES:
Feasibility of infusing MSCs into men with localized prostate cancer who plan to undergo a prostatectomy. | Up to 3 years
  The percentage of screened subjects that agreed to receive a pre-prostatectomy infusion of MSCs at the pre-specified time point and subsequently undergo a radical prostatectomy.
Determine the proportion of MSC to recipient DNA in the peripheral blood | Up to 3 years
  Proportion of MSC to recipient DNA is calculated by number of MSCs over the number of recipient DNA ([number of MSC]/[number of recipient DNA]) in the peripheral blood.
Determine the proportion of MSC to recipient DNA within the seminal vesicle. | Up to 3 years
  Proportion of MSC to recipient DNA is calculated by number of MSCs over the number of recipient DNA ([number of MSC]/[number of recipient DNA]) in the seminal vesicle.
Changes in the Sexual Health Inventory for Men (SHIM) survey post-prostatectomy. | Up to 3 years
  The SHIM is a measure of sexual function with a score ranging from 1 (severe erectile dysfunction) to 25 (normal function). Participants are required to have a score of >=17 to be eligible for the study.
Change in urinary function as assessed by the Expanded Prostate Cancer Index Composite (EPIC) survey post-prostatectomy | Baseline to Up to 3 years
  Change in total urinary function score (possible score range from 5-51) on the EPIC survey.
Change in bowel habits as assessed by the Expanded Prostate Cancer Index Composite (EPIC) survey post-prostatectomy | Baseline to Up to 3 years
  Change in total bowel habits score (possible score range from 8-62) on the EPIC survey.
Change in sexual function as assessed by the Expanded Prostate Cancer Index Composite (EPIC) survey post-prostatectomy | Baseline to Up to 3 years
  Change in total sexual function score (possible score range from 10-61) on the EPIC survey.
Change in hormonal function as assessed by the Expanded Prostate Cancer Index Composite (EPIC) survey post-prostatectomy | Baseline to Up to 3 years
  Change in total hormonal function score (possible score range from 5-49) on the EPIC survey.
Change in overall satisfaction as assessed by the Expanded Prostate Cancer Index Composite (EPIC) survey post-prostatectomy | Baseline to Up to 3 years
  Change in overall satisfaction score (possible score range from 1-5) on the EPIC survey with a higher score reflecting higher overall satisfaction.
Safety as assessed by number of participants experiencing adverse events | Up to 3 years
  Number of participants experiencing adverse events as defined by the revised National Cancer Institute Common Toxicity Criteria (NCI CTC), version 4.0 published 14 June 2010.
Safety as assessed by number of participants experiencing serious adverse events | Up to 3 years
  Number of participants experiencing serious adverse events as defined by the revised National Cancer Institute Common Toxicity Criteria (NCI CTC), version 4.0 published 14 June 2010.
Safety as assessed by number of participants experiencing treatment-related adverse events | Up to 3 years
  Number of participants experiencing treatment-related adverse events as defined by the revised National Cancer Institute Common Toxicity Criteria (NCI CTC), version 4.0 published 14 June 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235